CLINICAL TRIAL: NCT04222517
Title: The Use of Local Hemostatic in Patients With Large Incisional Hernias: Randomized Controlled Trial Study
Brief Title: The Use of Local Hemostatic in Patients With Large Incisional Hernias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nijznevartovsk County Clinical Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2020-01-04; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Hernia, Ventral
Keywords: hernia
MeSH Terms: conditions — Hernia, Ventral; Hernia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standart sublay retromuscular technique (Experimental): Apply standard intervention (sublay retromuscular)
  Interventions: Procedure: Incisional hernia repair by the mesh implant in sublay retromusuclar position
- Standart sublay retromuscular technique with Hemoblock (Experimental): Local hemostatic Hemoblock is used in retro-muscular and subcutaneous spaces
  Interventions: Procedure: Incisional hernia repair by the mesh implant in sublay retromusuclar position with using a local hemostatic Hemoblock

INTERVENTIONS:
Procedure: Incisional hernia repair by the mesh implant in sublay retromusuclar position — Incisional hernia repair using mesh prolene implant in sublay retromuscular position. Dissect the posterior rectus sheets, suture them continuously, formed a retromuscular space in which the standard prolene mesh implant is installed. Perform hemostasis. Install the drainage tube into the retromuscular space.
  After that, the anterior rectus sheets were sutured, hemostasis was performed, a drainage tube was installed in the subcutaneous tissue. Drainage tubes were connected to the UnoVac vacuum aspiration system (Unomedical, Denmark).
  Arms: Standart sublay retromuscular technique
Procedure: Incisional hernia repair by the mesh implant in sublay retromusuclar position with using a local hemostatic Hemoblock — Incisional hernia repair using mesh prolene implant in sublay retromuscular position. Dissect the posterior rectus sheets, suture them continuously, formed a retromuscular space in which the standard prolene mesh implant is installed. Perform hemostasis. Install the drainage tube into the retromuscular space. Used a local hemostatic Hemoblock 15 ml in this space.
  After that, the anterior rectus sheets were sutured, hemostasis was performed, a drainage tube was installed in the subcutaneous tissue. Used a local hemostatic Hemoblock 15 ml in subcutaneus space. Drainage tubes were connected to the UnoVac vacuum aspiration system (Unomedical, Denmark).
  Arms: Standart sublay retromuscular technique with Hemoblock

SUMMARY:
Design of a simple blind randomized controlled trial study. Large incisional hernia repair with use of local hemostatic Hemoblock

DETAILED DESCRIPTION:
Design of a simple blind randomized controlled trial study. The total number of subjects was 66. In the main group (A) - 33, in the other group (B) - 33. Operation - sublay retromuscular using prolene mesh implant. In group A Hemoblock 15 ml in the retromuscular and 15 ml in the subcutaneous spaces were used. Wounds were drained by vacuum-suction drainage. Postoperative monitoring of early ultrasound examinations on the 3rd, 7th, 10th, 12th, 15th, 18th, 21st, 25th, 28th, 30th days after drainage removal.

In group B were used a standard intervention (sublay retromuscular).

ELIGIBILITY:
Inclusion Criteria:

1. ASA I, II, III
2. the absence of oncological pathology
3. consent to participate in the study
4. Large incisional hernia (hernial defect ≥10 cm in diameter and/or area of hernial defect ≥100 cm2) according to the classification of EHS, 2009 (W3); age 25-75 years

Exclusion Criteria:

1. age older than 75 years
2. decompensated concomitant pathology, ASA≥IV
3. patient refusal to participate in the study

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2020-01-04 (Actual)

PRIMARY OUTCOMES:
drainage duration | from 1 to 6 days after operation
  Duration of drainage in days
the amount of the exudate from post-op wound | from 1 to 6 days after operation
  How many ml is exudate from the wound
the ultrasound changes of fluid collections in the postoperative wound | on the 3rd, 7th, 10th, 12th, 15th, 18th, 21st, 25th, 28th, 30th days after drainage removal.
  volume of the fluid collections in the post-op wound after drains removal
the number of necessary punctures of the postoperative wound | up to 30 days after drains removal
  How many punctures need to treatment fluid collections
amount of seromas | up to 30 days after drains removal
  use Morales-Conde classification
other postoperative wound complications | up to 30 days after drains removal
  such as SSI, thromboembolism, therapeutic complications
white blood cell count in exudate from post-op wound | from 1 to 6 days after operation
  The number of leukocytes
the number of lymphocytes in exudate from post-op wound | from 1 to 6 days after operation
  The number of lymphocytes
the amount of C-RP in exudate from post-op wound | from 1 to 6 days after operation
  The number of C-RP
the amount of Albuminum in exudate from post-op wound | from 1 to 6 days after operation
  The number of Albuminum

SECONDARY OUTCOMES:
Lenght of the Hospital stay | from 4 to 18 days
  Days
post-operative pain scores using numerical rating on Visual Analogue Scale (VAS) | Ten days after surgery twice a day (at 06:00 AM and at 06:00 PM).
  Ten days after surgery twice a day (at 06:00 AM and at 06:00 PM). A ten-point scale, where 0 points - no pain and 10 points - unbearable pain
The concentration of NSAD in mg of applied analgesics | up to 7-10 days after surgery
  NSAD (Ketoprofen)
The concentration of Tramadol in mg of applied analgesics | up to 7-10 days after surgery
  Tramadol
The concentration of Trimeperidine in mg of applied analgesics | up to 7-10 days after surgery
  Trimeperidine
Duration of use NSAD in days | up to 7-10 days after surgery
  NSAD (Ketoprofen)
Duration of use Tramadol in days | up to 7-10 days after surgery
  Tramadol
Duration of use Trimeperidine in days | up to 7-10 days after surgery
  Trimeperidine

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Kolyadko, Principal Investigator — Omsk state Medical Univesity
Locations (1):
- Nijnevartovsk Clinical County Hospital, Nizhnevartovsk, Russia

IPD SHARING:
Plan to Share IPD: No